CLINICAL TRIAL: NCT01219595
Title: Cranberry Proanthocyanidins for Modification of Intestinal E. Coli Flora and Prevention of Urinary Tract Infections in UTI-Susceptible Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Ocean Spray Cranberries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: H-2010-0107
Record Dates: First submitted 2010-10-08; First posted 2010-10-13 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Urinary Tract Infection
Keywords: Urinary Tract Infection; UTI
MeSH Terms: conditions — Urinary Tract Infections | interventions — Observation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Part 1 (Active Comparator): 1 serving (1/3 cup; 42 g) of sweetened, dried cranberries each day for two weeks.
  Interventions: Other: Sweetened, dried cranberries
- No treatment (Other): 20 non-UTI susceptible women will be enrolled to collect data on the types of E. coli flora present in non-UTI women.
  Interventions: Other: Observation
- Part 2A (Active Comparator): 1 serving (1/3 cup; 42 g) of sweetened, dried cranberries each day for three separate, two-week periods. Each two week period will be separated by a two-week interval.
  Interventions: Other: Sweetened, dried cranberries
- Part 2B (Placebo Comparator): 1 serving (1/3 cup; 42 g) of strawberry fruit pieces each day for three separate, two-week periods. Each two week period will be separated by a two-week interval.
  Interventions: Other: Strawberry Fruit Pieces
- Part 3A (Active Comparator): 1 serving (1/3 cup; 42 g) of sweetened, dried cranberries each day for one 4-week period.
  Interventions: Other: Sweetened, dried cranberries
- Part 3B (Placebo Comparator): 1 serving (1/3 cup; 42 g) of strawberry fruit pieces each day for one 4-week period.
  Interventions: Other: Strawberry Fruit Pieces

INTERVENTIONS:
Other: Sweetened, dried cranberries — Women in Arm 1 will consume one serving (1/3 cup; 42 g) of sweetened, dried cranberries each day for two weeks.
  Arms: Part 1; Part 2A; Part 3A
Other: Strawberry Fruit Pieces — 1 serving (1/3 cup; 42 g) of strawberry fruit pieces each day for three separate, two-week periods. Each two week period will be separated by a two-week interval.
  Arms: Part 2B; Part 3B
Other: Sweetened, dried cranberries — 1 serving (1/3 cup; 42 g) of sweetened, dried cranberries each day for three separate, two-week periods. Each two week period will be separated by a two-week interval.
  Arms: Part 1; Part 2A; Part 3A
Other: Sweetened, dried cranberries — 1 serving (1/3 cup; 42 g) of sweetened, dried cranberries each day for one 4-week period.
  Arms: Part 1; Part 2A; Part 3A
Other: Strawberry Fruit Pieces — 1 serving (1/3 cup; 42 g) of strawberry fruit pieces each day for one 4-week period.
  Arms: Part 2B; Part 3B
Other: Observation — Subjects in the non-UTI susceptible group will have one visit where one vaginal and one rectal swab will be collected.
  Arms: No treatment

SUMMARY:
The purpose of the research is to determine if eating sweetened, dried cranberries or strawberry fruit pieces will increase the types of different E. coli bacteria in the intestines which may reduce the likelihood of a major, or highly harmful urinary type of bacteria which cause urinary tract infections in susceptible women.

DETAILED DESCRIPTION:
This is a research study about the number and types of bacteria that cause urinary tract infections (E. coli strains) that are present in the intestine. The bacteria will be collected and analyzed before and after eating either sweetened, dried cranberries or strawberry fruit pieces. This study will help us learn more about whether or not the components of consumed sweetened, dried cranberries or strawberry fruit pieces reduce the numbers of harmful E. coli bacteria in the vaginal and intestinal tracts, thereby reducing the number of urinary tract infections among women.

ELIGIBILITY:
Inclusion Criteria:

* Women, ages 18-65
* History of recurrent urinary tract infections defined as three in the past year, or two in the last six months
* Subjects must be willing to follow the study protocol that includes consuming the mandatory daily dose of cranberries or strawberry fruit pieces and traveling to the UWHC Urology clinic for scheduled rectal and vaginal swab procedures.

The non-UTI-susceptible group will include women ages 18-65 with no history of recurrent UTI's as defined above.

Exclusion Criteria:

Women who:

* Are pregnant
* Have an immune compromising disease
* Have diabetes
* Have kidney stones
* Have chronic bowel inflammatory disease
* Have known allergies to cranberries, strawberries, elderberries, or wheat fiber

Non-UTI-susceptible group will include women ages 18-65 with no history of recurrent UTI's as defined above.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2010-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Pre-treatment heterogeneity or prevalence | Day 1 - prior to start of study treatment
  1) Prevalence or heterogeneity of E. coli strains in UTI susceptible women pre-treatment
Post-treatment heterogeneity | 2 weeks, 1 month, or 3 months
  2) a change in the heterogeneity of strains post treatment
Patient acceptance of study regimen | 2 weeks, 1 month, or 3 months
  3) patient acceptance of the study regimen
Maintenance of heterogeneity in the intestinal flora | Approximately 3 months
  To determine whether a shift towards strain heterogeneity in the intestinal flora can be maintained over a three month period.
Measure Effects of sweetened, dried cranberries on E. coli clonotypes over three two-week exposures | Approximately 3 months
  Measure effects of sweetened, dried cranberries on E. coli clonotypes over three two-week exposures
Measure effects of sweetened, dried cranberries on E. coli clonotypes over one 4-week exposure | 2 weeks, 1 month, or 3 months
  Measure effects of sweetened, dried cranberries on E. coli clonotypes over one 4-week exposure
Measure the UTI recurrence | 2 weeks, 1 month, or 3 months
  Measure the UTI recurrence after 6 months from the beginning of the study.
Comparison of sweetened dried cranberries to a placebo group | 2 weeks, 1 month, or 3 months
  Comparison of sweetened dried cranberries to a placebo group (strawberry fruit pieces)

CONTACTS AND LOCATIONS:
Overall Officials: Walter Hopkins, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States